CLINICAL TRIAL: NCT00196534
Title: A Comparative Evaluation of Human Thrombin Versus Bovine Thrombin in Achieving Hemostasis in Patients Undergoing Cardiovascular, Neurologic (Spine) and General Surgery Procedures.
Brief Title: A Study to Compare Human Thrombin Against Bovine Thrombin in Its Ability to Stop Bleeding After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 400-04-005
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular, Neurologic (Spine), and General Surgery
MeSH Terms: conditions — Neurologic Manifestations | interventions — Thrombin

INTERVENTIONS:
Drug: Human Thrombin
Drug: Bovine Thrombin

SUMMARY:
The purpose of this study is to see if Human Thrombin is as effective as Bovine Thrombin in stopping surgical bleeding within 10 minutes of application.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, of any race, 18 years or older.
* Patients who have at least one bleeding site within the operative field that is mild (oozing or capillary bleeding) to moderate (gradual or steady bleeding) in intensity and which cannot be managed by surgical modalities because they are ineffective or impractical (Change 15, Amend 1).
* Patients scheduled for any of the following elective surgical procedures:

  1. Cardiovascular Procedures - aortic surgery such as aneurysmectomy, aneurysmoplasty, aneurysmorrhaphy, aneurysmotomy and bypass procedures involving the aorta; major coronary bypass procedures including primary bypass surgery and re-do procedures. Peripheral vascular procedures to include femoral-popliteal bypass, femoral-femoral bypass, or other peripheral vascular procedures requiring vessel grafting with native or prosthetic grafts including Polytetrafluoroethylene (PTFE) grafts; carotid endarterectomies. The sternum is excluded as a Target Site. Bleeding sites evaluated during these procedures may include soft tissues (e.g. mammary bed, retroperitoneal fat/connective tissues and adhesions) and needle hole bleeding of prosthetic graft material (Change 6, Amend 1).
  2. Neurosurgical (spine) Procedures- primary lumbar laminectomy and laminectomy with fusion (fusion must be done after the time to hemostasis assessment). Re-do laminectomy, removal of tumors/lesions during laminectomy, cervical, or thoracic laminectomy procedures will be excluded. Bleeding sites evaluated may include periosteum, bone marrow, venous plexus (Change 7, Amend 1).
  3. General Surgery or Post-Traumatic (hemodynamically stable and non-coagulopathic) procedures: bowel and colon resections, retroperitoneal dissections/resections, and procedures involving the resection of any solid abdominal organ such as a splenectomy, liver resection, nephrectomy, splenorrhaphy, and pancreatectomy. Bleeding sites evaluated may include soft tissues (e.g. bowel mesentery, adhesions, lymph node beds, sacral venous plexus, etc.) and parenchymal organ bleeds (cut surface of resected liver, spleen, etc., excluding cut surface of kidney) (Amendment #2, Change 44). Bowel anastomoses sites will not be included (Change 8, Amend 1).
* Patient, or the patient's legally authorized representative, must provide legally effective informed consent prior to any participation in the study. (Amendment #2, Change 41)

Exclusion Criteria:

* Patients with bleeding diathesis, pathologic coagulopathy, systemic disorders, or autoimmune, immunodeficiency diseases or any other disorder that may interfere with hemostasis.
* Patients who have had a pre-operative laboratory finding that was considered clinically significant (as determined by the Investigator) for CBC (HCT, Hgb, white blood cell differential, platelet count, and Red Blood Cell (RBC) indices (MCH, MCV, MCHC)), prothrombin time (PT), or activated partial thromboplastin time (aPTT).
* Patients who have used anticoagulant, antiplatelet or nonsteroidal anti-inflammatory analgesic (NSAID) within 5 days prior to surgery (the use of ASA or aprotinin is permitted).
* Patients with known antibodies to bovine thrombin preparations.
* Patients receiving an organ transplant (liver, heart, kidney, etc.).
* Patients who are morbidly obese (Body Mass Index > 35).
* Patients with acute or chronic liver failure (Amendment #2, Change 42).
* Patients with all severe (brisk or forceful) bleeding site(s).
* Patients with an ongoing infection at the operative site.
* Patients who are known alcohol and/or drug abusers.
* Female patients who are pregnant or nursing.
* Patients who have uncontrolled diabetes mellitus (blood glucose levels >400 mg/dl) as determined by the Investigator based on medical history (Change 14, Admin. Change 2).
* Patients who have participated in another investigational drug or device research within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304
Dates: Start 2004-11; Study Completion 2006-07

PRIMARY OUTCOMES:
Success in achieving hemostasis.

SECONDARY OUTCOMES:
Success in achieving hemostasis after application
Estimated intraoperative blood loss
Procedure duration
Time in specialty units
Length of hospital stay
Incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Northwest NeuroSpecialists, PPLC, Tucson, Arizona
  - Vacular Surgery Associates, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - Ochsner Clinic, New Orleans, Louisiana
  - Union Memorial Hospital, Baltimore, Maryland
  - Borgess Research Institute, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebrask Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - Scott and White Hospital, Temple, Texas
  - Neurospine Center of Wisconsin, Appleton, Wisconsin

REFERENCES:
- [Derived] Doria C, Fischer CP, Wood CG, Li PM, Marra S, Hart J. Phase 3, randomized, double-blind study of plasma-derived human thrombin versus bovine thrombin in achieving hemostasis in patients undergoing surgery. Curr Med Res Opin. 2008 Mar;24(3):785-94. doi: 10.1185/030079908X273426. Epub 2008 Jan 31. PMID 18241525